CLINICAL TRIAL: NCT03049839
Title: Evaluation of a Community Health Program for the Prevention of Type 2 Diabetes and Other Cardio-metabolic Risk Factors in Adults: Districts of Barranquilla and Bogota, Colombia - January 2017 - December 2019
Acronym: PREDICOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad del Norte (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 55657
Record Dates: First submitted 2016-10-21; First posted 2017-02-10 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention_ structured (Experimental): One year Structured intervention program for members of high-risk group (People with glucose intolerance in the OGTT and FINDRISC score ≥12 points) 10 educational group sessions where they will receive information to change lifestyle (1 per 1.5 month)
  Interventions: Behavioral: Intervention_ S
- Intervention_ Informative (Experimental): Program information intervention for the group with moderate risk. One year Informative intervention program (People with normotolerant or impaired fasting glucose in the OGTT and FINDRISC score ≥12 points).
  There is a single group session where they receive information to prevent cardiomatabolic risk factors
  Interventions: Behavioral: Intervention_ I
- Intervention_ Communitarian (Experimental): One year, Intervention program at Community level. People with a FINDRISC less than 12 points.
  Campaigns are carried out at the community level with different strategies (leaflets, booklets) to prevent cardiomatabolic risk factors
  Interventions: Behavioral: Intervention_ C

INTERVENTIONS:
Behavioral: Intervention_ S — One year Structured intervention program for members of high-risk group (Subjects with FINDRISC score ≥12 points and impaired glucose tolerance (IGT))
  Other Names: LIP_Structures
  Arms: Intervention_ structured
Behavioral: Intervention_ I — One year Informative intervention program for members of moderate risk group (People with normotolerant or impaired fasting glucose in the OGTT and a FINDRISC score ≥12 points)
  Other Names: LIP_Informative
  Arms: Intervention_ Informative
Behavioral: Intervention_ C — One year, Intervention program at Community level. People with a FINDRISC less than 12 points
  Other Names: LIP_Communitarian
  Arms: Intervention_ Communitarian

SUMMARY:
The main aim of this study is to evaluate the feasibility and effectiveness of a program for modifying lifestyles for diabetes prevention type 2 and control cardio-metabolic risk factors in adults with different categories of risk from the primary health care strategy.

The project will show the effect of these interventions for the first time in people With different risk of developing type 2 diabetes throughout the life in populations living in Colombia Located in 2 different cities, one of them in the interior of the country (districts of Bogota) and another in the north coast (districts of Barranquilla) .

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) and type 2 diabetes (T2D) are currently the public health problems fastest growing globally. According to the International Diabetes Federation (IDF) is estimated to have diabetes approximately 382 million people in the world. It is shown that early interventions in lifestyle can reduce the burden of type 2 diabetes and factors of cardiovascular modifiable risk.

This is an intervention study in cluster. 36-month integrated into 4 phases:

1. Design and adaptation of educational intervention
2. Population Screening
3. Stepwise intervention program
4. Evaluation results.

For population screening test FINDRISC validated for the Latin American population will be employed and a score of 12 will be considered as a cutoff to all who have a score equal to or greater than 12 (moderate or high risk) they perform a test oral glucose tolerance (OGTT) according to the results 3 groups will be established

* High risk group: Subjects with FINDRISC score ≥12 and impaired glucose tolerance (IGT)
* Moderate risk group: Subjects with FINDRISC score ≥12 and impaired fasting glucose or norm tolerant
* Low risk group: Subjects with FINDRISC score <12.

Intervention program: One year of duration, 3 types of programs are established.

* Lifestyle Intervention program_ Communitarian: Intervention program at Community level with Low risk group.
* Lifestyle Intervention program_ Informative: Program information intervention for the group with moderate risk.
* Lifestyle Intervention program_ structured: intervention program for members of high-risk group.

An evaluation of the different variables are studied at baseline and the final of the intervention in the three groups established.

ELIGIBILITY:
Inclusion Criteria:

* People over age 30 years, residents within the perimeter of the conglomerate in the districts of Barranquilla and Bogota
* Wishing to participate and sign informed consent

Exclusion Criteria:

* DT2 known and / or treated
* History of diseases or events that prevent their participation
* Neurological disability that does not allow you to make own decisions
* Pregnant women

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of body weight average at year-end structured intervention compared with the baseline. | 12 Months
  Reduction of body weight in kilograms

SECONDARY OUTCOMES:
Reduction of fasting glucose level at year-end intervention program (all groups) compared with baseline. | 12 Months
  Reduction of fasting glucose level in mg/dl
Reduction of 2-hour glucose level at year-end structured and informative intervention program compared with baseline. | 12 Months
  Reduction of 2-hour glucose level in mg/dl
Reduced of waist circumference average at year-end structured intervention program compared with baseline. | 12 Months
  Reduction of waist circumference in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Tania Acosta, MD, MPH, Principal Investigator — Universidad del Norte; Pablo Achner, MD, ENDOCRINOLOGIST, Principal Investigator — ASOCIACIÓN COLOMBIANA DE DIABETES
Locations (2):
- Colombia (2):
  - Universidad Del Norte, Barranquilla
  - Asociación Colombiana de Diabetes, Bogotá

IPD SHARING:
Plan to Share IPD: No